CLINICAL TRIAL: NCT01708967
Title: One-time Spray of Epinephrine (1cc) Plus 4% Lidocaine (4cc) is Sufficient Pretreatment Method for the Preparation of Transnasal Endoscopy
Brief Title: Trial of New Pretreatment Method in Transnasal Endoscopy
Acronym: RTNPMTNE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Ki Tae Suk, doctor, assistant professor, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OTSMVSSCM
Record Dates: First submitted 2012-10-16; First posted 2012-10-17 (Estimated); Results first posted 2014-03-13 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-01

CONDITIONS: Pretreatment Method of Transnasal Endoscopy
Keywords: transnasal endoscopy; pretreatment method

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Catheter-free method (Experimental): We explored success rate, side effects, and vital signs in patients with catether-free method.
  Intervention: one-time spray of epinephrine (1cc) plus 4% lidocaine (4cc)
  Interventions: Procedure: pretreatment method for transnasal endoscopy
- Catheter insertion method (Experimental): We explored success rate, side effects, and vital signs in patients with catether insertion method : use both spray and catheter
  Interventions: Procedure: pretreatment method for transnasal endoscopy

INTERVENTIONS:
Procedure: pretreatment method for transnasal endoscopy — Catheter-free method : The patient then takes simethicone (10cc). After that, the nasal cavity is sprayed with epinephrine (1cc) and lidocaine HCL (4%, 4cc).
  Catheter inesertion method: After preparation steps the same as in the 'catheter-free' method, a 14 Fr. flexible catheter is coated with 2% lidocaine HCL gel and 8% lidocaine HCL spray. After that, the catheter is inserted into the patient's nasal cavity, and maintained about 1 minute for anesthesia. A 16 Fr. catheter is prepared by the same method with as the 14Fr. catheter. After the 14 Fr. cathter has been removed from the patient's nasal cavity, the 16 Fr. catheter is inserted into the patient's nasal cavity.
  Other Names: Catheter-free method/Cathter insertion method

SUMMARY:
This study designed for compare efficacy of following two anesthetic method for transnasal endoscopy

* "Catheter-free method"
* "Catheter-insertion method"

DETAILED DESCRIPTION:
1. Check of the medical history (both method)

   1. underlying systemic disease
   2. drug allergy
   3. anticoagulant or antiplatelet use
2. Premedication (both method)

   1. taking premedication contain dimethylpolysiloxane, pronase, sodium bicarbonate for improved endoscopic visualization
   2. spraying naphazolin acetate into nasal cavity for decrease secretion
3. Different anesthetic method for transnasal endoscopy

   1. "Catheter-free method" : spraying epinephrine into nasal cavity
   2. "Catheter-insertion method" : spraying both epinephrine and lidocaine into nasal cavity

ELIGIBILITY:
Inclusion Criteria:

* Routine check-up patients

Exclusion Criteria:

* nasal operation, an allergy, a possibility of hemorrhage

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ki Tae Suk, M.D.,Ph.D., Principal Investigator — Department of Internal Medicine, Hallym University Chuncheon Sacred Heart Hospital
Locations (1):
- Department of Internal Medicine, Hallym University Chuncheon Sacred Heart Hospital, Chuncheon, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Catheter-free Method: We explored success rate, side effects, and vital signs in patients with one-time spray method.
  Intervention: one-time spray of epinephrine (1cc) plus 4% lidocaine (4cc)
  pretreatment method for transnasal endoscopy : one-time spray method : patients are given simethicone (5cc) and lidocaine (2%, 10cc). After that, epinephrine (1cc) and lidocaine (2%, 3cc) are injected in both nose and mouth. Lastly, buscopan Intra Muscular (IM) is injected.
  spray+catheter method: patients are given simethicone (10cc). Next, epinephrine and lidocaine (4%, 4cc) are injected in both nose and mouth. Following this step, benoxinate hydrochloride (5cc) is inhaled by the patients. Subsequently, the patients are catheterized for 10 minutes using the 7Fr. Nelaton catheter. Finally, buscopan IM is injected.
- Catheter-insertion Method: We explored success rate, side effects, and vital signs in patients with spray+catheter method.
  Intervention: use both spray and catheter
  pretreatment method for transnasal endoscopy : one-time spray method : patients are given simethicone (5cc) and lidocaine (2%, 10cc). After that, epinephrine (1cc) and lidocaine (2%, 3cc) are injected in both nose and mouth. Lastly, buscopan Intra Muscular (IM) is injected.
  spray+catheter method: patients are given simethicone (10cc). Next, epinephrine and lidocaine (4%, 4cc) are injected in both nose and mouth. Following this step, benoxinate hydrochloride (5cc) is inhaled by the patients. Subsequently, the patients are catheterized for 10 minutes using the 7Fr. Nelaton catheter. Finally, buscopan IM is injected.
Period: Overall Study
Arm/Group | Catheter-free Method | Catheter-insertion Method
Started | 50 | 50
Completed | 50 | 43
Not Completed | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Catheter-free Method: We explored success rate, side effects, and vital signs in patients with one-time spray method.
  Intervention: one-time spray of epinephrine (1cc) plus 4% lidocaine (4cc)
- Catheter-insertion Method: We explored success rate, side effects, and vital signs in patients with spray+catheter method.
  Intervention: use both spray and catheter
- Total: Total of all reporting groups
Arm/Group | Catheter-free Method | Catheter-insertion Method | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 37 | 76
  >=65 years | 11 | 13 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (10.8) | 59.7 (12.3) | 59.00 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 52
  Male | 25 | 23 | 48
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 50 | 50 | 100

OUTCOME MEASURES:

1. Secondary Outcome: Vital Signs
Description: Blood pressure, heart rate, and O2 saturation were assessed.
Time Frame: before, during, and after transnasal endoscopy
Reporting Status: Not Posted

2. Other Pre Specified Outcome: Satisfaction
Description: Patients were asked to score how well they felt during endoscopy using a visual analog scale; they were also asked whether they would accept one-time spray method or spray+catheter method in the future if necessary.
Time Frame: after transnasal endoscopy
Reporting Status: Not Posted

3. Primary Outcome: Success Rate of Transnasal Endoscopy
Description: We difine the success of transnasal endoscopy as follows: the pateint underwent transnasal endoscopy without signicant complaint nor side effects.
  We difine the failure of transnasal endoscopy as follows: the patient cannot tolerate insertion of the endoscope; the patient presents side effects such as epistaxis, pain, or a decrease in O2 saturation; and the endoscope cannot pass through the nasal or oral cavity.
Time Frame: During transnasal endoscopy, up to 1 hours
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Catheter-free Method | Catheter-insertion Method
Number analyzed (Participants) | 50 | 43
percentage of Participants | 88 [80 to 96] | 88 [80 to 96]

ADVERSE EVENTS:
Arm/Group | Catheter-free Method | Catheter-insertion Method
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/43
Other Adverse Events (participants affected / at risk) | 0/50 | 0/43

LIMITATIONS AND CAVEATS:
A limitation of this study was the small number of patients; n = 93 is insufficient to conclusively generalize the efficiency of the catheter-free method.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other